CLINICAL TRIAL: NCT00237848
Title: D-Serine Augmentation of Cognitive Retraining in Schizophrenia
Brief Title: D-Serine for Enhancing Cognitive Retraining for the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other); Donaghue Foundation (Unknown); US Department of Veterans Affairs (U.S. Federal Agency); VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RPA/020/03; 1R01DA022495 (NIH); 103T-363
Record Dates: First submitted 2005-09-13; First posted 2005-10-12 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Drug: D-serine
Behavioral: Cognitive retraining

SUMMARY:
This study will examine the effectiveness of D-serine in increasing and sustaining the benefits of cognitive retraining in people with schizophrenia.

DETAILED DESCRIPTION:
This study is based on the hypothesis that by increasing NMDA receptor function in the brain and thereby increasing the capacity of the brain to both form new connections and strengthen existing connections, schizophrenic patients may derive both greater and sustained benefit from cognitive retraining.

Patients with schizophrenia or schizoaffective disorder who are currently receiving antipsychotic medication will be randomly assigned in a double-blind manner to receive either D-serine (30 mg/kg) or placebo in addition to cognitive rehabilitation or a non-interactive placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Clinically stable
* Treated with antipsychotic medications for at least 6 months in the past, and on a stable dose of the same antipsychotic medication over the past month
* Not pregnant or lactating

Exclusion Criteria:

* Other current or past DSM-IV Axis I diagnosis
* Calgary Depression scale score >10 or Simpson-Angus Rating Scale score > 20
* Currently treated with clozapine, lamotrigine or carbamazepine, or defined as treatment refractory
* Substance abuse or dependence within the past 3 months, except for nicotine
* Wechsler Adult Intelligence Scale-Revised score < 70
* Significant recent (within past 3 months) risk of committing suicide
* Abnormal thyroid function tests within the last 6 months
* Previous treatment with D-serine
* History of evidence of a medical or neurological condition that would expose the subject to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the trial
* Clinically significant abnormal laboratory test results at screening
* ECT treatment within the past two months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2005-02

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS)
Wisconsin Card Sorting Test (WCST)
Hopkins Verbal Learning Test
Spatial working memory task

SECONDARY OUTCOMES:
Heinrichs-Carpenter Quality of Life Scale
Neurocognitive training tasks
Functional assessments

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C. D'Souza, MD, Principal Investigator — Yale University
Locations (1):
- National Institute of Mental Health and Neurosciences, Bangalore, Karnataka, India

REFERENCES:
- [Background] Tsai GE, Yang P, Chung LC, Tsai IC, Tsai CW, Coyle JT. D-serine added to clozapine for the treatment of schizophrenia. Am J Psychiatry. 1999 Nov;156(11):1822-5. doi: 10.1176/ajp.156.11.1822. PMID 10553752
- [Background] Tsai G, Yang P, Chung LC, Lange N, Coyle JT. D-serine added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 1998 Dec 1;44(11):1081-9. doi: 10.1016/s0006-3223(98)00279-0. PMID 9836012
- [Background] Heresco-Levy U, Javitt DC, Ebstein R, Vass A, Lichtenberg P, Bar G, Catinari S, Ermilov M. D-serine efficacy as add-on pharmacotherapy to risperidone and olanzapine for treatment-refractory schizophrenia. Biol Psychiatry. 2005 Mar 15;57(6):577-85. doi: 10.1016/j.biopsych.2004.12.037. PMID 15780844